CLINICAL TRIAL: NCT03669458
Title: A Non-RandomizeD FEasibility Trial of the Spur SystEm for the Treatment of Lesions in the InfraPoplitEal ArteRy
Brief Title: Feasibility Clinical Trial Using the SPUR System to Demonstrate Safety and Efficacy.
Acronym: DEEPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ReFlow Medical, Inc. (Industry)
Collaborators: Syntropic Corelab (Unknown); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: CP-001
Record Dates: First submitted 2018-08-29; First posted 2018-09-13 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: A minimum of 10 patients will be enrolled for treatment of BTK disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Arm 1: BTK intervention with SPUR/DCB (Experimental): Below the knee peripheral intervention using SPUR/DCB.
  Interventions: Device: Below the Knee peripheral intervention
- Arm 2: BTK intervention using SPUR Only (Experimental): Below the knee peripheral intervention using SPUR only.
  Interventions: Device: Below the Knee peripheral intervention
- ARM 3: BTK intervention using DCB Only (Experimental): Below the knee peripheral intervention using DCB only.
  Interventions: Device: Below the Knee peripheral intervention

INTERVENTIONS:
Device: Below the Knee peripheral intervention — Treatment of infrapopliteal disease using SPUR/DCB, SPUR only and DCB alone
  Other Names: DCB Treatment; SPUR with DCB treatment

SUMMARY:
To evaluate the safety and effectiveness of the Spur System in a patient population with infrapopliteal artery disease (tibioperoneal, anterior/posterior tibial and peritoneal arteries) when used in conjunction with substance/drug coated balloons.

DETAILED DESCRIPTION:
The objective of this study is to perform a prospective, multi-center (min 2 sites), non-randomized study to evaluate the safety and efficacy of the Spur system and compare treatments arms (if applicable) in treating subjects with infrapopliteal disease who are at risk for amputation.

The study protocol will ensure consistency in performing the procedure, patient management and results of the procedure. Safety and efficacy will be evaluated during index procedure through one (1) year follow up

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to provide informed consent and able to comply with the study protocol.
* Peripheral arterial disease that can be treated using PTA.
* Life expectancy >1 year in the investigator's opinion
* Male or non-pregnant female > 18 years of age
* Patent inflow artery
* Target vessel(s) reconstitutes(s) at or above the ankle, excluding the dorsalis pedis and the calcaneal branch of the posterior tibial artery
* Target lesion starts at or below 3 cm below the tibial plateau as measured by angiography
* Target vessel for Spur device is ≥ 3.5 mm (4mm); ≥ 2.5 mm (3mm) in diameter by visual estimate.
* Lesion(s) must be able to be treated with a minimum of one Spur or PTA or DCB product.
* Infrapopliteal lesion(s) that are located in either the left or right leg Infrapopliteal artery(s) may be treated with only one modality per artery: DCB, Spur or Spur/DCB.
* Arterial length/diameter and quantity must be able to be treated with DCB or Spur or Spur/DCB
* The treated segment is defined as the total length of artery treated with PTA.
* The cumulative treated segment of infrapopliteal artery(s) must be ≤34.0 cm.
* Lesions in the treated segment may be continuous or may have gaps present between stenosis or occlusions
* Patient has Rutherford Classification of 3-5.
* Successful pre-dilatation of the target lesion.
* Iliac, SFA and popliteal inflow lesions can be treated during the same procedure using standard angioplasty and/or approved device. These inflow lesions must be treated first, prior to consideration of treatment of infrapopliteal lesions.
* The patient can be enrolled if the inflow lesions have acceptable angiographic results (must have <30% residual stenosis and no evidence of embolization or flow limiting dissection)

Exclusion Criteria:

* Subject unwilling or unlikely to comply with the appropriate follow up time for the duration of the study
* Prior stent(s) or bypass surgery within the target vessel(s)
* Target lesion is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion.
* Previous treatment failure of inflow arteries (Iliac, SFA and popliteal) which required a surgical procedure.
* Previous PTA of the target vessel within 30 day prior to index procedure
* Angiographic evidence of thrombus within target limb.
* Subject has an active infection of the foot, including pus or wet gangrene that is not controlled at the time of the procedure.
* Planned major (above the ankle) amputation of the target limb
* Recent MI or stroke < 30 days prior to the index procedure.
* Heart failure with Ejection Fraction < 30%
* Impaired renal function (GFR <30 mL/min) and patients on dialysis
* Subject with vasculitis, systemic Lupus Erythematosus or Polymyalgia Rheumatica.
* Patient receiving systemic corticosteroid therapy.
* Inability to tolerate concomitant antiplatelet and oral anticoagulation therapy.
* Known allergies or sensitivities to heparin, aspirin (ASA), other anticoagulant therapies which could not be substituted, and/or paclitaxel or an allergy to contrast media that cannot be adequately pre-treated prior to the index procedure.
* The patient is currently enrolled in another investigational device or drug trial that is interfering with the endpoints of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Demonstrate binary arterial flow at 6 months | 6 months
  The primary effectiveness endpoint assess arterial flow using duplex ultrasound at 6 months post procedure.

SECONDARY OUTCOMES:
MALE | 30 days
  The secondary safety endpoint assess Freedom from Major Adverse Limb events (MALE) at 30 days
All cause perioperative death (30 days) | 30 days
  The secondary safety endpoint assess all-cause perioperative death (POD) at 30 days

OTHER OUTCOMES:
Device and procedure related death through 30 days post procedure. | 30 days
  The safety endpoint assess freedom from device and procedure-related death through 30 days post-procedure and freedom from target limb major amputation
Clinically driven target lesion revascularization through 12 months post procedure. | 12 months
  The safety endpoint assess clinically driven target lesion revascularization through 12 months post procedure
Freedom from major target amputation through 30 days from the device or procedure | 30 days
  The safety endpoint from freedom of major target amputation.

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Mustapha, MD, Principal Investigator — Advanced Cardiac & Vascular Centers
Locations (1):
- Instituto Nacional de la Diabetes (INDEN), Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No
All data need to be analyzed